CLINICAL TRIAL: NCT00137163
Title: Evaluation of Dermafill Dressing for Autogenous Skin Donor Sites
Brief Title: Evaluation of Dermafill Dressing for Donor Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Institute of Surgical Research (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-04-026
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2008-07-28 (Estimated); Status verified 2008-07

CONDITIONS: Burns
Keywords: burns; donor site care; Dermafill dressing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dermafill Dressing

SUMMARY:
The purpose of the study is to compare one type of dressing against the current standard dressing that is used to cover the unburned area of the skin where a piece of skin is removed to cover another part of the body that was burned.

Hypothesis: The mean healing time for wounds treated with the Dermafill dressing will be less than the mean healing time for wounds treated with Xeroform dressing.

DETAILED DESCRIPTION:
At the time of the procedure, donor sites that are symmetrical in size and shape will be selected. The donor sites will be harvested. Once the grafts have been harvested, the wounds will be randomized for treatment using either the Dermafill dressing or Xeroform. The wound dressings will then be observed at least once a day beginning post op day 2/48hours after surgery until healed, which is defined as 90% or more of the wound surface is confluently re-epithelized.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older; male or female.
* Burn wounds less than 30% of total body surface area (TBSA) with no systemic abnormalities
* Burns do not involve the harvesting area
* Burn wounds require excision and grafting of sufficient extent to justify two donor sites of equal and symmetrical size on non-dependent body surface areas
* Scheduled excision and grafting procedure is the first such operation for subject during this hospitalization
* Subject agrees to participate in follow-up evaluations

Exclusion Criteria:

* Critical illnesses requiring ventilator support, systemic infection or hemodynamic instability
* Major acute or chronic illnesses affecting wound healing (e.g. peripheral vascular disease, insulin dependent diabetes, blood clotting disorder)
* Subject receiving medications that inhibit/compromise wound healing (e.g. anticoagulants, antiplatelet drugs, oral steroids). The use of anticoagulants does not include deep venous thrombosis (DVT) prophylaxis.
* Cellulitis or other infection of potential donor site
* Previously harvested donor site
* Subjects with greater than 30% TBSA burns
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17
Dates: Start 2005-03; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Pain will be less or equal to with the Dermafill dressing as compared with Xeroform
Cosmetic effect of healing at post surgery day 30-60 will be equal or less with Dermafill as compared with Xeroform

SECONDARY OUTCOMES:
Infections associated with donor sites will be equal to or less with Dermafill as compared with Xeroform

CONTACTS AND LOCATIONS:
Overall Officials: Michael Albrecht, MD, Principal Investigator — US Army Institute of Surgical Research
Locations (1):
- US Army Institute of Surgical Research, Fort Sam Houston, Texas, United States